CLINICAL TRIAL: NCT03851796
Title: The Role of Parents in Adolescent Obesity Treatment: Randomized Control Trial of TEENS+
Brief Title: Parent Involvement in Adolescent Obesity Treatment
Acronym: TEENS+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of North Carolina (Other); University of Tennessee (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20014304; R01HD095910-01A1 (NIH)
Record Dates: First submitted 2018-12-12; First posted 2019-02-22 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Obesity
Keywords: Pediatric Obesity; Lifestyle Intervention; Family-based Intervention; Motivational Interviewing
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessors and the PI will be blind to treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEENS+Parents as Coaches (Active Comparator): Parents are taught strategies to support and facilitate child weight management via family-based change. Each visit includes group psychoeducation and discussion, focused on strategies to facilitate healthy weight management in their child(ren). Topics include role modeling, strategies for healthy lifestyle changes, and how to be a coach to your teen. They receive personalized feedback throughout the program.
  All adolescents participate in a group-based empirically supported behavioral weight management treatment, that includes dietary and physical activity goals, and instructions to self-monitor key information. Adolescents will receive training in core behavioral weight loss strategies (e.g. goal setting, stimulus control) and techniques to help them achieve these goals. They also receive personalized feedback throughout the program.
  Interventions: Behavioral: TEENS+Parents as Coaches
- TEENS+Parent Weight Loss (Active Comparator): Parents are given a weight loss goal of 1-2 lbs/week, and specific calorie and fat prescriptions, PA goals, and instructions to self-monitor key information. Parents receive training in core behavioral weight loss strategies (e.g. goal setting, stimulus control) and techniques to help them achieve these goals. They also receive personalized feedback throughout the program.
  All adolescents participate in a group-based empirically supported behavioral weight management treatment, that includes dietary and physical activity goals, and instructions to self-monitor key information. Adolescents receive training in core behavioral weight loss strategies (e.g. goal setting, stimulus control) and techniques to help them achieve these goals. They also receive personalized feedback throughout the program.
  Interventions: Behavioral: TEENS+Parent Weight Loss

INTERVENTIONS:
Behavioral: TEENS+Parents as Coaches — Parents as Coaches teaches parenting strategies to facilitate healthy weight loss in adolescent children; adolescents are in a group based behavioral weight management treatment.
  Other Names: Parents as Champions for TEENS (PACT)
  Arms: TEENS+Parents as Coaches
Behavioral: TEENS+Parent Weight Loss — Parent Weight loss teaches core behavioral weight loss strategies and techniques for parent weight loss; adolescents are in a group based behavioral weight management treatment.
  Other Names: Healthy You!
  Arms: TEENS+Parent Weight Loss

SUMMARY:
A randomized control trial to compare the efficacy of two distinct parent treatments on weight loss maintenance for adolescents with obesity participating in a lifestyle intervention including nutrition education, exercise and behavioral support.

Funding support from NIH via 1R01HD095910

DETAILED DESCRIPTION:
Investigators will recruit adolescents with overweight or obesity (BMI>85th percentile) and a parent (BMI > 25 kg/m2). Families will participate in one of two 4-month treatments: 1) TEENS+ Parents as Coaches (PAC), engaging parents as helpers in their child's weight management, or 2) TEENS+ Parent Weight Loss (PWL), engaging parents in their own weight management. All adolescents will participate in TEENS+, which includes behavioral support, nutrition education, and supervised physical activity.

For adolescents, the intervention will consist of weekly behavioral weight management group sessions and weekly 1 hour exercise sessions. Each adolescent also has a monthly individual session with a behavior coach. Parent groups meet weekly for 1 hour according to treatment arm (PAC or PWL). All PWL sessions are separate from their adolescent. Bi-weekly sessions in the PAC arm are combined with parents and adolescent. Assessments will consist of anthropometric measures, psychological surveys and dietary and PA evaluations. Assessments will be completed at baseline, 2 months, 4 months (post-test), 8 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

Adolescent Inclusion Criteria:

* BMI ≥ 85th percentile for age and gender according to the CDC Growth Charts
* Age 12 to 16
* Must reside with the primary participating parent

Parent Inclusion Criteria:

* ≥18
* BMI ≥ 25 kg/m2
* Must reside with the adolescent

Exclusion Criteria:

Adolescent Exclusion Criteria:

* Non-English speaking
* Medical condition(s) that may be associated with unintentional weight change
* Diabetes mellitus
* Use of oral glucocorticoids, atypical antipsychotics, weight loss medications, or an investigational medication within 3 months of study participation
* Use of a GLP-1 within 6 months of study participation
* Use of Depo-Provera within 6 months of study participation
* Medical condition(s) that may be negatively impacted by exercise
* Psychiatric, cognitive, physical or developmental conditions that would impair the ability to complete assessments, participate in a group, or conduct physical activity
* Reports of compensatory behaviors in the past 3 months
* Current pregnancy or plan to become pregnant during study period
* Previous participation in HM20010365, HM20003076, HM20005235 or HM20014304
* Current participation in another weight loss program
* Personal history of weight loss surgery
* Severe depression
* Clinically significant eating disorder
* Change in dose of metformin, tricyclic antidepressants, selective serotonin uptake inhibitors, or stimulant medications within 3 months of study participation
* Admission to a psychiatric hospital within the past year

Parent Exclusion Criteria:

* Non-English speaking
* Medical condition(s) that may be associated with unintentional weight change
* Use of oral glucocorticoids, atypical antipsychotics, weight loss medications, or an investigational medication within 3 months of study participation
* Use of a GLP-1 within 6 months of study participation with no T2D diagnosis; if T2D diagnosis, change in dose GLP-1 within 3 months of study participation
* Use of Depo-Provera within 6 months of study participation
* Psychiatric, cognitive, physical or developmental conditions that would impair the ability to complete assessments, participate in a group, or conduct physical activity
* Reports of compensatory behaviors in the past 3 months
* Current pregnancy, lactation, less than 6 months post-partum, or plan to become pregnant during study period
* Previous participation in HM20010365, HM20003076, HM20005235 or HM20014304
* Current participation in another weight loss program
* Personal history of weight loss surgery
* Severe depression
* Clinically significant eating disorder
* Change in dose of diabetes medications, tricyclic antidepressants, selective serotonin uptake inhibitors, or stimulant medications within 3 months of study participation
* Admission to a psychiatric hospital within the past year

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 418 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2024-10-26 (Actual); Study Completion 2024-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie K Bean, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at VCU Healthy Lifestyles Center, Henrico, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown KL, LaRose JG, Raynor HA, Gorin AA, Thornton LM, Farthing S, Tatum K, Bean MK. Study design and rationale for TEENS+REACH: Evaluating ripple effects of a family-based lifestyle intervention to untreated family members. Contemp Clin Trials Commun. 2024 Feb 15;38:101276. doi: 10.1016/j.conctc.2024.101276. eCollection 2024 Apr. PMID 38404649
- [Derived] Bean MK, LaRose JG, Wickham EP 3rd, Raynor HA, Caccavale L, Evans RK, Thornton LM, Farthing S, Mendoza A, Mazzeo SE. The role of parents in behavioral treatment for adolescent obesity: design and rationale for the TEENS+ randomized clinical trial. BMC Public Health. 2023 Aug 4;23(1):1484. doi: 10.1186/s12889-023-16421-0. PMID 37537548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the trial occurred from March 2019 through August 2023 with more strategized recruitment methods occurring 3-4 months prior to the start of each cohort. We implemented a comprehensive recruitment plan which included: establishing relationships with community practices for provider referrals; physician-endorsed letters; direct mail; social media and targeted digital ads; local newspaper/magazine/radio ads; flyers/posters in medical offices/hospital; listservs; community events.
Groups:
- Teens with parents in PAC: All adolescents participate in a group-based empirically supported behavioral weight management treatment, that includes dietary and physical activity goals, and instructions to self-monitor key information. Adolescents receive training in core behavioral weight loss strategies (e.g. goal setting, stimulus control) and techniques to help them achieve these goals. They receive personalized feedback throughout the program.
  These adolescents have a participating parent in the Parents as Coaches (PAC) treatment arm.
- Teens with parents in PWL: All adolescents participate in a group-based empirically supported behavioral weight management treatment, that includes dietary and physical activity goals, and instructions to self-monitor key information. Adolescents receive training in core behavioral weight loss strategies (e.g. goal setting, stimulus control) and techniques to help them achieve these goals. They receive personalized feedback throughout the program.
  These adolescents have a participating parent in the Parent Weight Loss (PWL) treatment arm.
- Parents as Coaches (PAC): Parents are taught strategies to support and facilitate child weight management via family-based change. Each visit includes group psychoeducation and discussion, focused on strategies to facilitate healthy weight management in their child(ren). Topics include role modeling, strategies for healthy lifestyle changes, and how to be a coach to your teen. They receive personalized feedback throughout the program.
- Parent Weight Loss (PWL): Parents are given a weight loss goal of 1-2 lbs/week, and specific calorie and fat prescriptions, PA goals, and instructions to self-monitor key information. Parents receive training in core behavioral weight loss strategies (e.g. goal setting, stimulus control) and techniques to help them achieve these goals. They receive personalized feedback throughout the program.
Period: Overall Study
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Started | 107 | 104 | 105 | 102
Completed | 86 | 94 | 84 | 92
Not Completed | 21 | 10 | 21 | 10

BASELINE CHARACTERISTICS:
Groups:
- Teens With Parents in PAC: All adolescents participate in a group-based empirically supported behavioral weight management treatment, that includes dietary and physical activity goals, and instructions to self-monitor key information. Adolescents receive training in core behavioral weight loss strategies (e.g. goal setting, stimulus control) and techniques to help them achieve these goals. They receive personalized feedback throughout the program.
- Total: Total of all reporting groups
Arm/Group | Teens With Parents in PAC | Teens With Parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL) | Total
Number analyzed (Participants) | 107 | 104 | 105 | 102 | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (1.3) | 13.54 (1.4) | 44.44 (6.8) | 43.87 (7.7) | 28.69 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 60 | 89 | 85 | 295
  Male | 46 | 44 | 16 | 17 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 5 | 4 | 29
  Not Hispanic or Latino | 95 | 95 | 99 | 97 | 386
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 5 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 53 | 43 | 51 | 44 | 191
  White | 43 | 39 | 46 | 46 | 174
  More than one race | 4 | 10 | 2 | 3 | 19
  Unknown or Not Reported | 2 | 7 | 1 | 6 | 16
Region of Enrollment [Number; unit: participants]
  United States | 107 | 104 | 105 | 102 | 418
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.27 (6.49) | 34.71 (6.97) | 36.02 (8.10) | 36.27 (7.75) | 35.31 (7.37)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI) Change
Description: Body Mass Index (BMI) change (kg/m2; adolescent) during the maintenance phase (4-month to 12-month).
Time Frame: 4 months to 12 month [follow up phase]
Population: Data presented includes the participants who completed body weight measurements at the respective time points [4 & 12m] and the change in BMI between the two time points.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Teens with parents in PAC | Teens with parents in PWL
Number analyzed (Participants) | 84 | 93
kg/m^2 | 1.51 (2.44) | 0.91 (2.27)

2. Primary Outcome: Body Mass Index
Description: National Health and Nutrition Examination Survey (NHANES) Anthropometry methods were used to measure height and weight to calculate Body Mass Index (BMI). At 0, 2, 4, 8, 12 months, trained staff measured adolescent height and weight (in light clothing and after a 12 hour fast) to the nearest 0.1cm and 0.1kg using a precision stadiometer and digital scale, respectively.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Data presented includes the participants who completed body weight measurements at the respective time points.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Teens with parents in PAC | Teens with parents in PWL
Number analyzed (Participants) | 107 | 104
kg/m^2
  Baseline | 34.27 (6.49) | 34.71 (6.97)
  2-month: number analyzed (Participants) | 103 | 99
  2-month | 33.58 (6.55) | 34.16 (7.03)
  4-month: number analyzed (Participants) | 99 | 97
  4-month | 33.21 (6.39) | 33.92 (7.13)
  8-month: number analyzed (Participants) | 91 | 93
  8-month | 33.66 (6.99) | 34.56 (7.49)
  12-month: number analyzed (Participants) | 86 | 94
  12-month | 34.09 (7.26) | 34.79 (7.51)

3. Secondary Outcome: Parent Weight
Description: Trained staff will measure weight (in light clothing and after a 12 hour fast) to the nearest 0.1kg using digital scale at baseline, 2-, 4-, 8- and 12-months.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Data presented includes the participants who completed body weight measurements at the respective time points.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 105 | 102
Kilograms
  Baseline | 99.18 (22.93) | 100.62 (26.17)
  2-month: number analyzed (Participants) | 101 | 97
  2-month | 97.39 (20.16) | 98.51 (26.17)
  4-month: number analyzed (Participants) | 97 | 94
  4-month | 98.50 (24.31) | 96.06 (24.65)
  8-month: number analyzed (Participants) | 91 | 91
  8-month | 97.29 (23.04) | 96.69 (25.37)
  12-month: number analyzed (Participants) | 84 | 87
  12-month | 95.97 (22.33) | 98.25 (25.74)

4. Secondary Outcome: Parent Weight Change
Description: Trained staff will measure weight (in light clothing and after a 12 hour fast) to the nearest 0.1kg using digital scale at baseline and 4-months. Weight change will be calculated from these values.
Time Frame: baseline to 4 month [intervention phase] and 4 month to 12 month [maintenance phase]
Population: Data presented includes the participants who completed body weight measurements at the respective time points ([0 & 4m] and [4 & 12m]) and the change in weight between the two time points.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 97 | 94
Kilograms
  0-4 month change | -1.20 (4.11) | -3.47 (4.51)
  4-12 month change: number analyzed (Participants) | 82 | 86
  4-12 month change | -0.32 (6.59) | 0.49 (1.76)

5. Secondary Outcome: Physical Activity
Description: Accelerometers were worn for 1 week by adolescents and parents for each assessment period (0, 4, 8, and 12 months) to assess adolescent and parent physical activity. Results represent total time (minutes/day) spent in moderate/vigorous activity (MVPA). Data reported is based off the average MVPA minutes per day of valid wear days.
Time Frame: Baseline, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 107 | 104 | 105 | 102
minutes per day
  Baseline: number analyzed (Participants) | 101 | 100 | 104 | 97
  Baseline | 11.99 (12.11) | 11.92 (11.75) | 21.05 (17.83) | 22.51 (18.54)
  4-month: number analyzed (Participants) | 85 | 79 | 88 | 81
  4-month | 12.03 (15.85) | 12.41 (12.35) | 19.75 (16.99) | 24.65 (18.46)
  8-month: number analyzed (Participants) | 77 | 73 | 81 | 77
  8-month | 10.78 (14.39) | 15.48 (13.74) | 19.09 (13.88) | 21.93 (17.69)
  12-month: number analyzed (Participants) | 69 | 67 | 70 | 71
  12-month | 9.83 (12.44) | 13.90 (16.14) | 17.99 (13.26) | 21.55 (21.14)

6. Secondary Outcome: Physical Activity Change
Description: To assess adolescent and parent physical activity change during the maintenance physical (post-intervention) phase of the program from 4-months to 12-months. Results represent the change in total time (minutes/day) spent in moderate/vigorous activity (MVPA).
Time Frame: 4-month to 12-month
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 67 | 61 | 67 | 67
minutes per day | -3.21 (14.05) | 3.24 (14.11) | -1.28 (15.77) | -3.68 (14.35)

7. Secondary Outcome: Physical Activity Energy Expenditure
Description: Accelerometers will be worn for 1 week by adolescents and parents for each assessment period (0, 4, 8, and 12 months) to assess adolescent and parent physical activity energy expenditure (EE). Results represent the average daily physical activity energy expenditure (kilocalories/day) estimated via accelerometer. Results are based off EE = (Metabolic Equivalent of Task [MET] value of activity x body weight kg x [minutes of activity/60]) with MET values of 2.5, 4, and 7 utilized for light, moderate, and vigorous activities, respectively.
Time Frame: Baseline, 4-, 8-, and 12-months
Population: Results include participants who met the minimum monitor wear time (3 weekdays and 1 weekend day) at the respective time point.
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 107 | 104 | 105 | 102
kilocalories per day
  Baseline: number analyzed (Participants) | 83 | 92 | 93 | 93
  Baseline | 915.73 (370.39) | 897.27 (385.31) | 1486.38 (448.30) | 1506.10 (546.61)
  4-month: number analyzed (Participants) | 56 | 52 | 75 | 69
  4-month | 815.05 (317.61) | 856.47 (303.50) | 1349.37 (357.90) | 1542.45 (583.33)
  8-month: number analyzed (Participants) | 54 | 45 | 71 | 60
  8-month | 872.27 (337.40) | 900.97 (347.12) | 1399.80 (394.07) | 1541.63 (618.11)
  12-month: number analyzed (Participants) | 49 | 48 | 58 | 60
  12-month | 832.10 (333.46) | 871.07 (317.98) | 1347.41 (389.41) | 1496.42 (575.02)

8. Secondary Outcome: Physical Activity Energy Expenditure Change
Description: To assess adolescent and parent physical activity energy expenditure change during the maintenance physical (post-intervention) phase of the program from 4-months to 12-months. Results represent the change in total kilocalories per day from physical activity.
Time Frame: 4-month to 12-month
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 37 | 33 | 50 | 53
kilocalories per day | 10.30 (298.35) | 67.74 (244.26) | 9.57 (352.50) | -36.39 (417.73)

9. Secondary Outcome: Dietary Intake
Description: Adolescent and parent participants completed a 3-day food record to track dietary intake for 2 weekdays and 1 weekend day in the week prior to their assessment (0, 4, 8, 12m). Recall data was entered the Nutrition Data System for Research Software (NDSR) by trained staff. Parent and adolescent average total energy intake (kilocalories/day) from the logged days is reported.
Time Frame: Baseline, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 107 | 104 | 105 | 102
kilocalories per day
  Baseline | 1830 (493) | 1807 (546) | 1699 (511) | 1817 (622)
  4-month: number analyzed (Participants) | 94 | 91 | 92 | 87
  4-month | 1539 (501) | 1502 (529) | 1491 (432) | 1451 (405)
  8-month: number analyzed (Participants) | 84 | 86 | 83 | 81
  8-month | 1478 (466) | 1510 (493) | 1463 (736) | 1516 (483)
  12-month: number analyzed (Participants) | 75 | 84 | 73 | 77
  12-month | 1587 (475) | 1611 (447) | 1499 (470) | 1593 (447)

10. Secondary Outcome: Home Food Environment
Description: The Home Food Inventory (HFI) was used to assess the availability of types of food in the home and calculate an overall obesogenic score. Scores range from 0-60, with high scores indicating a more obesogenic food environment.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 105 | 102
score on a scale
  Baseline | 22.16 (7.44) | 22.28 (8.24)
  2-month: number analyzed (Participants) | 100 | 93
  2-month | 15.89 (6.35) | 18.54 (7.42)
  4-month: number analyzed (Participants) | 95 | 90
  4-month | 15.97 (6.81) | 17.09 (7.26)
  8-month: number analyzed (Participants) | 89 | 87
  8-month | 16.84 (7.22) | 17.95 (7.57)
  12-month: number analyzed (Participants) | 81 | 87
  12-month | 17.81 (7.29) | 18.20 (7.92)

11. Secondary Outcome: Parent Reported Parenting Style
Description: The Parenting Styles and Dimension Questionnaire (PSDQ) was administered to parents to assess parent self-report of authoritative parenting style. Results reflect the participating parent's perception of their parenting style. Scores range from 1-5 with higher scoring indicating a greater frequency of authoritative parenting behaviors.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point for each participating child. Parents who participated with 2 children responded to this measure twice.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Questionnaires
Arm/Group | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 105 | 102
Number analyzed (Questionnaires) | 107 | 104
score on a scale
  Baseline | 4.08 (0.47) | 4.12 (0.50)
  2-month: number analyzed (Participants) | 102 | 95
  2-month: number analyzed (Questionnaires) | 104 | 97
  2-month | 4.07 (0.45) | 4.10 (0.49)
  4-month: number analyzed (Participants) | 96 | 91
  4-month: number analyzed (Questionnaires) | 98 | 93
  4-month | 4.12 (0.52) | 4.15 (0.52)
  8-month: number analyzed (Participants) | 89 | 87
  8-month: number analyzed (Questionnaires) | 89 | 89
  8-month | 4.13 (0.51) | 4.14 (0.42)
  12-month: number analyzed (Participants) | 83 | 87
  12-month: number analyzed (Questionnaires) | 83 | 89
  12-month | 4.12 (0.54) | 4.16 (0.49)

12. Secondary Outcome: Role Modeling
Description: At 0, 2, 4, 8, 12 months, adolescents will complete the Family Experiences Related to Food Questionnaire (FERFQ) is an 8 or 9-item measure (father and mother version, respectively) that will assess family commentary about weight and shape as well as family modeling of diet and weight concerns. Scores range from 1-5 with higher scores indicating more negative role modeling of dietary behaviors. Results reflect the adolescent's perception on their parent (mom or dad) participating in the study.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Teens with parents in PWL: All adolescents participate in a group-based empirically supported behavioral weight management treatment, that includes dietary and physical activity goals, and instructions to self-monitor key information. Adolescents receive training in core behavioral weight loss strategies (e.g. goal setting, stimulus control) and techniques to help them achieve these goals. They receive personalized feedback throughout the program.
Arm/Group | Teens with parents in PAC | Teens with parents in PWL
Number analyzed (Participants) | 107 | 104
score on a scale
  Baseline: number analyzed (Participants) | 106 | 102
  Baseline | 2.54 (0.77) | 2.57 (0.85)
  2-month: number analyzed (Participants) | 103 | 96
  2-month | 2.46 (0.68) | 2.52 (0.75)
  4-month: number analyzed (Participants) | 95 | 92
  4-month | 2.33 (0.72) | 2.46 (0.82)
  8-month: number analyzed (Participants) | 85 | 85
  8-month | 2.29 (0.75) | 2.53 (0.88)
  12-month: number analyzed (Participants) | 79 | 87
  12-month | 2.32 (0.67) | 2.46 (0.83)

13. Secondary Outcome: Restrictive Child Feeding Practices
Description: Parents will complete the Child Feeding Questionnaire (CFQ; Adolescent version) to assess restrictive feeding style. Scores range from 1-5 with higher scores indicating a greater degree of restrictive feeding practices.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Questionnaires
Arm/Group | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 105 | 102
Number analyzed (Questionnaires) | 107 | 104
score on a scale
  Baseline | 3.54 (0.86) | 3.64 (0.77)
  2-month: number analyzed (Participants) | 101 | 95
  2-month: number analyzed (Questionnaires) | 103 | 97
  2-month | 3.36 (0.77) | 3.34 (0.84)
  4-month: number analyzed (Participants) | 95 | 91
  4-month: number analyzed (Questionnaires) | 97 | 93
  4-month | 3.17 (3.17) | 3.23 (0.89)
  8-month: number analyzed (Participants) | 89 | 87
  8-month: number analyzed (Questionnaires) | 89 | 89
  8-month | 3.12 (0.89) | 3.35 (0.84)
  12-month: number analyzed (Participants) | 82 | 87
  12-month: number analyzed (Questionnaires) | 82 | 89
  12-month | 3.20 (0.89) | 3.09 (0.87)

14. Secondary Outcome: Overall Weight Control Practices
Description: Adolescents and parents will complete the Weight Control Strategies Scale (WCSS) which will assess the use of healthy weight control practices (e.g., dietary choices, self-monitoring, and physical activity) at 0, 2, 4, 8, 12 months. A total of 30 items are included in the measure, rated from 0-4. Total scores (ranging from 0-4) are calculated by averaging the scores of the 30 items. Higher scores indicate greater engagement in weight management behaviors.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 107 | 104 | 105 | 102
score on a scale
  Baseline: number analyzed (Participants) | 107 | 103 | 105 | 102
  Baseline | 1.23 (0.67) | 1.12 (0.59) | 1.35 (0.75) | 1.22 (0.58)
  2-month: number analyzed (Participants) | 103 | 95 | 100 | 95
  2-month | 2.25 (0.77) | 2.22 (0.72) | 1.87 (0.69) | 2.18 (0.58)
  4-month: number analyzed (Participants) | 96 | 92 | 95 | 91
  4-month | 2.11 (2.11) | 2.10 (0.78) | 1.80 (0.70) | 2.20 (0.72)
  8-month: number analyzed (Participants) | 87 | 89 | 89 | 87
  8-month | 1.76 (0.80) | 1.77 (0.74) | 1.58 (0.75) | 1.76 (0.69)
  12-month: number analyzed (Participants) | 80 | 91 | 81 | 87
  12-month | 1.69 (0.80) | 1.58 (0.75) | 1.64 (0.75) | 1.52 (0.67)

15. Secondary Outcome: Self Monitoring Weight Control Practices
Description: Adolescents and parents will complete the Weight Control Strategies Scale (WCSS) self-monitoring subscale which will assess the use of self-monitoring weight control practices at 0, 2, 4, 8, 12 months. A total of 7 items are included in the measure, rated from 0-4. Scores are calculated by averaging the scores of the 7 items. Higher scores indicate greater engagement in self-monitoring weight management behaviors.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 107 | 104 | 105 | 102
score on a scale
  Baseline: number analyzed (Participants) | 107 | 103 | 105 | 102
  Baseline | 0.61 (0.75) | 0.52 (0.64) | 0.76 (0.83) | 0.53 (0.66)
  2-month: number analyzed (Participants) | 103 | 95 | 100 | 95
  2-month | 2.29 (0.98) | 2.25 (1.01) | 1.31 (1.02) | 2.46 (0.63)
  4-month: number analyzed (Participants) | 96 | 92 | 95 | 91
  4-month | 1.88 (1.08) | 1.84 (1.03) | 1.21 (0.96) | 2.23 (1.08)
  8-month: number analyzed (Participants) | 87 | 89 | 89 | 87
  8-month | 1.23 (1.00) | 1.20 (0.97) | 1.08 (0.98) | 1.32 (0.95)
  12-month: number analyzed (Participants) | 80 | 91 | 81 | 87
  12-month | 1.21 (1.02) | 1.02 (0.85) | 1.10 (0.97) | 1.00 (0.81)

16. Secondary Outcome: Dietary Choices Weight Control Practices
Description: Adolescents and parents will complete the Weight Control Strategies Scale (WCSS) dietary choices subscale which will assess the use of dietary choice weight control practices at 0, 2, 4, 8, 12 months. A total of 10 items are included in the measure, rated from 0-4. Scores range from 0 to 4 and are calculated by averaging the scores of the 10 items. Higher scores indicate greater engagement in dietary choice weight management behaviors.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 107 | 104 | 105 | 102
score on a scale
  Baseline: number analyzed (Participants) | 104 | 103 | 105 | 102
  Baseline | 1.90 (0.76) | 1.84 (0.74) | 2.22 (0.74) | 2.27 (0.66)
  2-month: number analyzed (Participants) | 103 | 95 | 100 | 95
  2-month | 2.65 (0.76) | 2.65 (0.68) | 2.82 (0.61) | 2.65 (0.63)
  4-month: number analyzed (Participants) | 96 | 92 | 95 | 91
  4-month | 2.63 (0.77) | 2.59 (0.76) | 2.75 (0.65) | 2.71 (0.61)
  8-month: number analyzed (Participants) | 87 | 89 | 89 | 87
  8-month | 2.35 (0.75) | 2.42 (0.71) | 2.46 (0.84) | 2.51 (0.62)
  12-month: number analyzed (Participants) | 80 | 91 | 81 | 87
  12-month | 2.23 (0.84) | 2.23 (0.79) | 2.51 (0.71) | 2.42 (0.66)

17. Secondary Outcome: Physical Activity Weight Control Practices
Description: Adolescents and parents will complete the Weight Control Strategies Scale (WCSS) physical activity subscale which will assess the use of physical activity weight control practices at 0, 2, 4, 8, 12 months. A total of 6 items are included in the measure, rated from 0-4. Scores range from 0 to 4 and are calculated by averaging the scores of the 6 items. Higher scores indicate greater engagement in physical activity weight management behaviors.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 107 | 104 | 105 | 102
score on a scale
  Baseline: number analyzed (Participants) | 107 | 103 | 105 | 102
  Baseline | 1.09 (0.96) | 0.91 (0.82) | 1.13 (1.06) | 0.86 (0.86)
  2-month: number analyzed (Participants) | 103 | 95 | 100 | 95
  2-month | 1.95 (1.00) | 1.88 (0.97) | 1.44 (1.05) | 1.68 (0.90)
  4-month: number analyzed (Participants) | 96 | 92 | 95 | 91
  4-month | 1.79 (1.14) | 1.81 (1.03) | 1.45 (0.99) | 1.78 (1.03)
  8-month: number analyzed (Participants) | 87 | 89 | 89 | 87
  8-month | 1.60 (1.14) | 1.60 (1.02) | 1.24 (1.00) | 1.34 (1.00)
  12-month: number analyzed (Participants) | 80 | 91 | 81 | 87
  12-month | 1.51 (1.02) | 1.46 (1.07) | 1.28 (1.09) | 1.11 (1.04)

18. Secondary Outcome: Psychological Coping Weight Control Practices
Description: Adolescents and parents will complete the Weight Control Strategies Scale (WCSS) psychological coping subscale which will assess the use of psychological coping weight control practices at 0, 2, 4, 8, 12 months. A total of 7 items are included in the measure, rated from 0-4. Scores range from 0 to 4 and are calculated by averaging the scores of the 7 items. Higher scores indicate greater engagement in psychological coping weight management behaviors.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 107 | 104 | 105 | 102
score on a scale
  Baseline: number analyzed (Participants) | 107 | 103 | 105 | 102
  Baseline | 1.31 (0.87) | 1.21 (0.82) | 1.28 (0.90) | 1.20 (0.80)
  2-month: number analyzed (Participants) | 103 | 95 | 100 | 95
  2-month | 2.12 (0.96) | 2.09 (0.86) | 1.92 (0.86) | 1.94 (0.73)
  4-month: number analyzed (Participants) | 96 | 92 | 95 | 91
  4-month | 2.15 (0.86) | 2.15 (0.88) | 1.78 (0.90) | 2.08 (0.83)
  8-month: number analyzed (Participants) | 87 | 89 | 89 | 87
  8-month | 1.84 (1.00) | 1.84 (0.93) | 1.53 (0.90) | 1.88 (0.84)
  12-month: number analyzed (Participants) | 80 | 91 | 81 | 87
  12-month | 1.82 (0.91) | 1.64 (0.92) | 1.65 (0.91) | 1.55 (0.89)

19. Secondary Outcome: Adolescent Reported Responsiveness Parenting Style
Description: The Authoritative Parenting Index (API) was used to assess adolescent-report of responsiveness parenting style and will be administered at 0, 2, 4, 8, 12 months. Scores range from 9-36 with higher scores indicating greater perceived responsiveness from the parent. Results reflect the adolescent's perception on the parent (mom or dad) participating in the study.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL
Number analyzed (Participants) | 107 | 104
score on a scale
  Baseline: number analyzed (Participants) | 103 | 97
  Baseline | 27.59 (5.52) | 28.09 (4.90)
  2-month: number analyzed (Participants) | 102 | 91
  2-month | 28.00 (5.66) | 28.84 (4.86)
  4-month: number analyzed (Participants) | 93 | 92
  4-month | 28.84 (5.15) | 29.12 (5.27)
  8-month: number analyzed (Participants) | 85 | 89
  8-month | 28.52 (5.64) | 28.67 (5.81)
  12-month: number analyzed (Participants) | 81 | 90
  12-month | 28.58 (5.32) | 28.10 (5.84)

20. Secondary Outcome: Adolescent Reported Demandingness Parenting Style
Description: The Authoritative Parenting Index (API) was used to assess adolescent-report of demandingness parenting style and will be administered at 0, 2, 4, 8, 12 months. Scores range from 7-28 with higher scores indicating greater perceived demandingness from the parent. Results reflect the adolescent's perception on their parent (mom or dad) participating in the study.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL
Number analyzed (Participants) | 107 | 104
score on a scale
  Baseline: number analyzed (Participants) | 103 | 97
  Baseline | 21.78 (4.07) | 21.59 (4.21)
  2-month: number analyzed (Participants) | 102 | 91
  2-month | 22.11 (4.16) | 21.87 (3.97)
  4-month: number analyzed (Participants) | 93 | 92
  4-month | 22.31 (4.29) | 21.75 (3.86)
  8-month: number analyzed (Participants) | 85 | 89
  8-month | 22.18 (4.16) | 22.04 (4.10)
  12-month: number analyzed (Participants) | 81 | 90
  12-month | 21.70 (4.58) | 21.40 (4.43)

21. Secondary Outcome: Adolescent Reported Authoritative Parenting Style
Description: The Authoritative Parenting Index (API) was used to assess adolescent-report of authoritative parenting style and was administered at 0, 2, 4, 8, 12 months. Scores range from 16-64 with higher scores indicating the adolescent perceives their parent to have a higher level of authoritative parenting behavior. Results reflect the adolescent's perception on their parent (mom or dad) participating in the study.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL
Number analyzed (Participants) | 107 | 104
score on a scale
  Baseline: number analyzed (Participants) | 103 | 97
  Baseline | 49.37 (7.62) | 49.68 (7.12)
  2-month: number analyzed (Participants) | 102 | 91
  2-month | 50.11 (8.01) | 50.70 (7.15)
  4-month: number analyzed (Participants) | 93 | 92
  4-month | 51.15 (8.00) | 50.87 (7.46)
  8-month: number analyzed (Participants) | 85 | 89
  8-month | 50.69 (8.06) | 50.72 (8.47)
  12-month: number analyzed (Participants) | 81 | 90
  12-month | 50.28 (8.58) | 49.50 (8.75)

22. Secondary Outcome: Home Exercise Environment
Description: The Exercise Environment Questionnaire (EEQ) assessed the availability of types exercise equipment in the home. Measures will be completed at 0, 4, 8, 12 months. Scores are calculated by summing responses. Scores range from 0-39 with higher scores indicating more exercise equipment in the home.
Time Frame: Baseline, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 105 | 102
score on a scale
  Baseline | 11.51 (5.51) | 11.11 (4.80)
  4-month: number analyzed (Participants) | 95 | 90
  4-month | 13.66 (5.35) | 12.74 (4.74)
  8-month: number analyzed (Participants) | 89 | 87
  8-month | 13.02 (6.36) | 12.23 (4.90)
  12-month: number analyzed (Participants) | 81 | 87
  12-month | 14.15 (5.31) | 13.33 (5.03)

23. Secondary Outcome: Monitoring Child Feeding Practices
Description: Parents will complete the Child Feeding Questionnaire (CFQ; Adolescent version) to assess monitoring feeding style. Scores range from 1-5 with higher scores indicating a greater degree of monitoring feeding practices.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Questionnaires
Arm/Group | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 105 | 102
Number analyzed (Questionnaires) | 107 | 104
score on a scale
  Baseline | 3.30 (0.99) | 3.21 (1.06)
  2-month: number analyzed (Participants) | 101 | 95
  2-month: number analyzed (Questionnaires) | 103 | 97
  2-month | 3.77 (0.94) | 3.41 (0.96)
  4-month: number analyzed (Participants) | 95 | 91
  4-month: number analyzed (Questionnaires) | 97 | 93
  4-month | 3.55 (1.04) | 3.25 (1.08)
  8-month: number analyzed (Participants) | 89 | 87
  8-month: number analyzed (Questionnaires) | 89 | 89
  8-month | 3.35 (1.09) | 3.21 (0.95)
  12-month: number analyzed (Participants) | 82 | 87
  12-month: number analyzed (Questionnaires) | 82 | 89
  12-month | 3.32 (1.04) | 3.08 (1.04)

24. Other Pre Specified Outcome: Autonomy Support
Description: At 0, 2, 4, 8, 12 months, adolescents will complete the Perceived Parental Autonomy Support Scale (P-PASS) to assess adolescent perception of 1) autonomy-supportive parenting behaviors and 2) controlling parenting behaviors. Items are rated on a 7-point Likert scale from 1-7. The average score across all items is calculated. Higher scores indicate a greater perception of parental autonomy support. Lower scores indicate less support and more controlling behaviors.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL
Number analyzed (Participants) | 107 | 104
score on a scale
  Baseline: number analyzed (Participants) | 94 | 93
  Baseline | 2.82 (4.01) | 3.00 (4.13)
  2-month: number analyzed (Participants) | 92 | 84
  2-month | 2.82 (4.00) | 2.75 (3.72)
  4-month: number analyzed (Participants) | 96 | 94
  4-month | 2.95 (3.87) | 3.02 (4.13)
  8-month: number analyzed (Participants) | 74 | 75
  8-month | 3.15 (4.61) | 3.00 (4.46)
  12-month: number analyzed (Participants) | 80 | 88
  12-month | 2.34 (3.58) | 3.31 (4.94)

25. Other Pre Specified Outcome: Parent Child Relationship
Description: The Conflict Behavior Questionnaire (CBQ; Parent and Adolescent Versions) will assess parent and adolescent report of parent-child relational factors at 0, 2, 4, 8, 12 mo. Scores range from 0-20. Higher score indicate more conflict between parent and child and lower scores indicating less conflict. Results reflect the adolescent's perception on their parent (mom or dad) participating in the study.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 107 | 104 | 105 | 102
score on a scale
  Baseline: number analyzed (Participants) | 94 | 93 | 95 | 93
  Baseline | 2.82 (4.01) | 3.00 (4.13) | 3.53 (4.66) | 3.82 (4.54)
  2-month: number analyzed (Participants) | 92 | 84 | 93 | 86
  2-month | 2.82 (4.00) | 2.75 (3.72) | 3.32 (4.34) | 3.47 (4.55)
  4-month: number analyzed (Participants) | 96 | 94 | 97 | 93
  4-month | 2.95 (3.87) | 3.02 (4.13) | 3.79 (4.44) | 3.31 (4.13)
  8-month: number analyzed (Participants) | 74 | 75 | 77 | 77
  8-month | 3.15 (4.61) | 3.00 (4.46) | 4.09 (5.03) | 3.36 (3.74)
  12-month: number analyzed (Participants) | 80 | 88 | 82 | 89
  12-month | 2.34 (3.58) | 3.31 (4.94) | 3.78 (4.82) | 3.47 (4.31)

26. Other Pre Specified Outcome: Parent Self-efficacy
Description: The Parent Efficacy for Child Healthy Weight Behavior (PECHWB) will assess parent self-efficacy in promoting healthy weight behaviors in their adolescents. Scores range from 0-100 with higher scores indicating higher self-efficacy.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
Number analyzed (Participants) | 42 | 39
score on a scale
  Baseline | 67.75 (23.24) | 66.58 (17.96)
  2-month: number analyzed (Participants) | 28 | 25
  2-month | 69.29 (18.33) | 62.44 (21.54)
  4-month: number analyzed (Participants) | 27 | 26
  4-month | 70.78 (16.99) | 59.42 (23.01)
  8-month: number analyzed (Participants) | 26 | 25
  8-month | 65.37 (17.86) | 62.11 (20.62)
  12-month: number analyzed (Participants) | 11 | 14
  12-month | 68.44 (20.34) | 57.59 (20.76)

27. Other Pre Specified Outcome: Social Support
Description: At 0, 2, 4, 8, 12 months, adolescents will complete family and friend social support scales from the Patient-based Assessment and Counseling for Physical Activity and Nutrition (PACE+) questionnaires to assess adolescent report of family and friend social support across 3 domains: 1) fruit and vegetable intake, 2) fat intake, and 3) physical activity. Scores range from 1-5 with higher indicating greater social support.
Time Frame: Baseline, 2-, 4-, 8-, and 12-months
Population: Results include participants who completed the measure at the respective time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens with parents in PAC | Teens with parents in PWL
Number analyzed (Participants) | 107 | 104
score on a scale
  Baseline: number analyzed (Participants) | 107 | 103
  Baseline | 3.04 (0.95) | 2.95 (0.78)
  2-month: number analyzed (Participants) | 103 | 95
  2-month | 3.58 (0.82) | 3.41 (0.86)
  4-month: number analyzed (Participants) | 96 | 95
  4-month | 3.44 (0.96) | 3.36 (0.99)
  8-month: number analyzed (Participants) | 87 | 89
  8-month | 3.21 (1.03) | 3.25 (0.92)
  12-month: number analyzed (Participants) | 81 | 91
  12-month | 3.05 (0.89) | 3.00 (1.07)

ADVERSE EVENTS:
Time Frame: 4-, 8-, and 12-months
Description: Adverse event information was collected at all post-intervention assessment time points (4, 8, and 12 months). Adverse events that were reported during active intervention 0-4 months, followed the same data collection protocol. A research coordinator collected information regarding the event onset date, ending date, specifics of the event (what was happening when it occurred, outcome, medications, follow up details).
Groups:
- Parent Weight Loss (PWL): family-based change. Each visit includes group psychoeducation and discussion, focused on strategies to facilitate healthy weight management in their child(ren). Topics include role modeling, strategies for healthy lifestyle changes, and how to be a coach to your teen. They receive personalized feedback throughout the program.
  Parents are given a weight loss goal of 1-2 lbs/week, and specific calorie and fat prescriptions, PA goals, and instructions to self-monitor key information. Parents receive training in core behavioral weight loss strategies (e.g. goal setting, stimulus control) and techniques to help them achieve these goals. They receive personalized feedback throughout the program.
Arm/Group | Teens With Parents in PAC | Teens With Parents in PWL | Parents as Coaches (PAC) | Parent Weight Loss (PWL)
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/104 | 0/105 | 0/102
Serious Adverse Events (participants affected / at risk) | 1/107 | 2/104 | 3/105 | 5/102
Other Adverse Events (participants affected / at risk) | 13/107 | 17/104 | 19/105 | 13/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teens With Parents in PAC (N=107) | Teens With Parents in PWL (N=104) | Parents as Coaches (PAC) (N=105) | Parent Weight Loss (PWL) (N=102)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Asthma attack requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Severe headache requiring hospitalization (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast reduction surgery requiring hospitalization (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Non-ST-elevation myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chemotherapy for Non-Hodgkin's lymphoma (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Side effects from therapy resulted in hospitalization
Psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gall bladder removal surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teens With Parents in PAC (N=107) | Teens With Parents in PWL (N=104) | Parents as Coaches (PAC) (N=105) | Parent Weight Loss (PWL) (N=102)
Muscle/Bone Injury (Musculoskeletal and connective tissue disorders) | 11 (14) | 13 (19) | 10 (11) | 7 (7)
Minor medical proceduree (Surgical and medical procedures) | 2 (2) | 4 (4) | 9 (10) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT03851796/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03851796/ICF_000.pdf